CLINICAL TRIAL: NCT05296876
Title: Multi-dimensional Evaluation of Carotid Artery Stenosis and Prediction of Brain Function After Endarterectomy by SSPC System
Brief Title: SSPC Evaluation on Carotid Artery Stenosis After Endarterectomy
Acronym: SSPC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Pudong Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ShanghaiPudong-SSPC
Record Dates: First submitted 2021-11-29; First posted 2022-03-25 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Carotid Stenosis; Carotid Artery Diseases; Carotid Artery Plaque
Keywords: carotid stenosis; carotid revascularization; symptoms; degree of stenosis; plaque; cerebral compensation
MeSH Terms: conditions — Carotid Stenosis; Carotid Artery Diseases; Plaque, Amyloid | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- carotid endarterectomy: Patients who are treated with CEA under SSPC evaluation
  Interventions: Procedure: Carotid endarterectomy (CEA)

INTERVENTIONS:
Procedure: Carotid endarterectomy (CEA) — Surgeons follow the contemporary guideline combined with their experience and preference in order to perform CEA for patients. All patients will be assessed by SSPC evaluation system before CEA. Patients will receive 100 mg of aspirin or 75 mg of clopidogrel daily starting from at least 72 h prior to the CEA procedure and continued receiving the medication indefinitely. General anesthesia is recommended for CEA and the type of CEA can be selected as conventional, eversion or a shunt or patch based on the discretion of the surgeon.

SUMMARY:
SSPC includes degree of Stenosis, Symptoms, Plaque stability and Compensation of the cerebral blood flow. SSPC, a comprehensive evaluation system on carotid artery stenosis, is established and advocated in this trial in order to make assessment on risk of carotid revascularization preoperatively and prediction of cerebral events postoperatively.

DETAILED DESCRIPTION:
Although, cerebral perfusion and collaterals recruitment are crucial and integral to current treatment and stroke prevention paradigms, most consensus recommendations do not include assessments of cerebral hemodynamics in their management algorithms and arbitrarily focus on symptoms and degree of stenosis.

Based on four aspects of SSPC multidimensional assessment and grading, through clinical data, specimen collection, image technology of the multi-disciplinary cross research, we initially to propose a more scientific evaluation system for the perioperative period of carotid revascularization, to reveal the scientific mechanism of brain function changes after carotid revascularization, and to establish a method for the evaluation of brain function after carotid revascularization in accordance with the characteristics of Chinese lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or patient's legal representative have been informed of the nature of the study, agrees to participate and has signed an Ethical Committee approved consent form
2. Unilateral or bilateral carotid artery stenosis diagnosed by ultrasound or CT angiography.
3. Complete revascularization followed by carotid endarterectomy or carotid artery stenting.

Exclusion Criteria:

1. Patients with carotid stenosis received best medicine therapy.
2. Patients for whom antiplatelet therapy, anticoagulants, medium contrast, or thrombolytic drugs are contraindicated.
3. Patient has bleeding diathesis, coagulopathy, known hypercoagulable condition or refuses blood transfusion
4. female patient with childbearing potential not taking adequate contraceptives or currently breastfeeding.
5. Life expectancy of less than twelve months.
6. Patient is currently participating in another investigational drug or device study that has not completed the entire follow up period.
7. Patient presenting one of the following comorbid conditions: hemodialysis, elevated creatine levels (> 2.5mg/dl), recent MI or ischemic stroke occurrence (both within 30 days).
8. Patient unwilling or unlikely to comply with Follow-Up schedule

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with carotid artery stenosis and fulfilled the above eligible criteria in tertiary medical centers in China, will be enrolled consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Stroke or TIA within 12 months | within 12 months post-procedure
  Number of participants with treatment-Stroke or TIA within 12 months
Immediate neurologic events within 24 hours | within 24 hours post-procedure
  Number of participants with treatment-immediate neurologic events including cerebral hyperperfusion syndrome, early-phase hypertension and cerebral hemorrhage within 24 hours
Cognition improvements | within 1, 3, 6, 12 months post-procedure
  Cognition improvements indicated by MMSE (Mini-mental State Examination) or MoCA (Montreal Cognitive Assessment) or Cantab (Cambridge Neuropsychological Test Automated Battery)

SECONDARY OUTCOMES:
Myocardial Infarction or death within 1 month | within 1 month post-procedure
  Number of participants with treatment-Myocardial Infarction or death within 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pudong Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No